CLINICAL TRIAL: NCT07312864
Title: A Clinical Trial Assessing the Safety, Tolerability, and Exploratory Efficacy of a Novel Bioartificial Liver Therapy in Patients With Liver Failure or Small-for-Size Syndrome
Brief Title: Safety and Tolerability Study of a Novel Bioartificial Liver in Liver Failure and Small-for-Size Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Li-Ying Sun, Director of Department of Critical Liver Diseases, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH20251124001
Record Dates: First submitted 2025-11-26; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Liver Failure; Small-for-Size Syndrome
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CiPS-BAL (Experimental): Chemically induced pluripotent stem cells biological Artificial Liver
  Interventions: Biological: Chemically induced pluripotent stem cells biological Artificial Liver

INTERVENTIONS:
Biological: Chemically induced pluripotent stem cells biological Artificial Liver — Participants will receive CiPS-BAL therapy, a novel bioartificial liver treatment that combines functional hepatocytes derived from chemically induced pluripotent stem cells (CiPS) with an extracorporeal bioartificial liver device . The CiPS-derived hepatocytes are cultured and induced in vitro under GMP conditions, then loaded into the BAL device for treatment. Therapy is administered via central venous access (e.g., femoral, internal jugular, or subclavian vein) for 4-8 hours per session. Each patient receives approximately 1.67 × 10^8 functional hepatocytes per kg of body weight, with treatment frequency and duration adjusted according to clinical response. Standard medical care for liver failure or small-for-size syndrome is provided alongside CiPS-BAL therapy. Patients are closely monitored for safety, tolerability, and changes in clinical and laboratory parameters.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of a novel bioartificial liver (CiPS-BAL) in patients with liver failure or small-for-size syndrome. The study will also collect preliminary data on clinical outcomes and laboratory parameters during treatment. The main questions it aims to answer are:

Is the novel bioartificial liver system safe and well tolerated in patients with liver failure or small-for-size syndrome?

What effects does the treatment have on liver function and other clinical and laboratory indicators?

Researchers will treat participants with the CiPS-BAL system, which uses hepatocytes derived from chemically induced pluripotent stem cells (CiPS) within a bioartificial liver device.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with liver failure (including acute, subacute/acute-on-chronic, and chronic liver failure) or small-for-size syndrome

Exclusion Criteria:

* Presence of severe extrahepatic systemic end-stage diseases

Uncontrollable infection or active bleeding

Pregnant or breastfeeding women

History of allergy or known severe hypersensitivity to CiPSC-derived cell products or blood products

Peripheral vascular collapse leading to inability to obtain venous access or collect blood

Unable or unwilling to provide informed consent or unable to comply with study requirements

Unwilling to receive CiPSC-based therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events and serious adverse events | From initiation of CiPS-BAL therapy through 12 months post-treatment (assessed at Day 7, Week 4, Week 12, Month 6, and Month 12)
  The number and proportion of participants experiencing treatment-emergent adverse events (AEs) and serious adverse events (SAEs) following CiPS-BAL therapy, including but not limited to fever, rash, chest tightness, palpitations, acute infusion reactions, immune rejection, infections, and local complications (e.g., hematoma, bleeding), and thrombosis.
  Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Survival and Liver Transplantation Rate | 7 days, 4 weeks, 12 weeks, 6 months, and 12 months after CiPS-BAL therapy.
  Overall survival of the patients and the proportion of participants who undergo liver transplantation during the study period.

SECONDARY OUTCOMES:
Change from baseline in Model for End-Stage Liver Disease (MELD) score | Baseline; 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after CiPS-BAL therapy
  The MELD score, a validated composite score based on serum bilirubin, international normalized ratio (INR), and serum creatinine, will be assessed at each follow-up visit.
  The outcome will be reported as the change from baseline in MELD score at each specified time point.
Glasgow Coma Scale (GCS) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
  GCS will be evaluated at each follow-up visit. The outcome will be reported as the change from baseline in GCS score.
SOFA Score | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
  SOFA score will be measured at each specified time point. The outcome will be reported as the change from baseline in SOFA score.
APACHE II Score | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
  APACHE II score will be assessed at scheduled time points. The outcome will be reported as the change from baseline.
Lactate | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
  Lactate levels will be measured from blood samples. The outcome will be reported as the change from baseline at each specified time point.
Alpha-Fetoprotein (AFP) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Ceruloplasmin | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Blood Ammonia | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
RBC (Red Blood Cell Count) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Hemoglobin (Hb) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
WBC (White Blood Cell Count) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Platelet Count (PLT) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
ALT (Alanine Aminotransferase) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
AST (Aspartate Aminotransferase) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Total Bilirubin (TBIL) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Direct Bilirubin (DBIL) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
ALP (Alkaline Phosphatase) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
BUN (Blood Urea Nitrogen) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Serum Creatinine (Scr) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Albumin (ALB) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Glucose (GLU) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Prothrombin Time (PT) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Prothrombin Activity (PTA) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
International Normalized Ratio (INR) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.
Activated Partial Thromboplastin Time (APTT) | 0.5-1 hour, 12 hours, 24 hours, Day 2, Day 3, Day 5, Day 7, Week 2, Week 4, Week 6, Week 12, Month 6, and Month 12 after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China